CLINICAL TRIAL: NCT01748097
Title: Phase III Study to Assess the Utility of a New Innovative Technique Using Intravenous Bicarbonate to Verify the Correct Position of Patients Scheduled for Intravenous Bicarbonate
Brief Title: Intravenous Bicarbonate To Verify The Correct Position of IV Catheters in Oncological Patients Oncological Patients Receiving Chemotherapy
Acronym: IVBICONCOL
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Netherlands: Ministry of Health, Welfare and Sports (Other Government)
Responsible Party: Principal Investigator, Dr. Ilan Keidan, director pediatric anesthesia, Sheba Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: IV BIC for IVONCOL
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Detection of the Correct Position of Intravenous Line
Keywords: infiltration; extravasation; sodium bicarbonate; capnography; end tidal carbon dioxide; chemotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV bicarbonate 4.2% 20 cc (Experimental): injecting 20cc 4.2% to a newly administered IV line
  Interventions: Drug: sodium bicarbonate 4.2%
- IV normal saline (Placebo Comparator): injecting 20 cc normal saline to a newly administered IV line

INTERVENTIONS:
Drug: sodium bicarbonate 4.2%
  Arms: IV bicarbonate 4.2% 20 cc

SUMMARY:
The investigators use bicarbonate injected to an intravenous line and the changes in the exhaled end-tidal carbon dioxide to verify whether the IV line is in the vein or surrounding tissue

DETAILED DESCRIPTION:
The method was proved useful in previous phase I, II studies. Now the investigators move on to assess the method in a phase III study in oncological patients.

each patients which will be subjected to intravenous chemotherapy will be eligible ( see also inclusion/exclusion criteria).

Once consent obtained the patient will have an IV line placed. each line placed will be categorized by the clinical team into 3 categories:

1. IV in place ready to use for chemotherapy ( good blood return)
2. Doubtful position ( no blood return/ little blood return bu flushes well).
3. IV not in place. Study design Category 1. IV bicarbonate 4.2% 20 cc and NS 20 cc in a randomized fashion Category 2. same as above Category 3. No injections

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 oncological disease requires intravenous chemotherapy

Exclusion Criteria:

* 1. refusal to participate 2. lung disease acute or chronic sPo2 < 92%, PaCO2 > 50 3. renal failure Creatinine > 2 mg% 4. metabolic alkalosis HCO3 > 30 meq/L 5. medication that affect bicarbonate levels: Bicarbonate, Diamox, Fusid 6. obesity BMI > 38 7. congestive heart failure EF < 40 % or clinical signs of congestive heart failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
change in exhaled end tidal co2 | 1-3 minutes
  the injection of bicarbonate in a vein cause a rapid and distinct change in exhaled end-tidal CO2

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Sheba Medical Center Oncology, Tel Litwinsky, Israel
  - Oncology Clinic, Tel Litwinsky